CLINICAL TRIAL: NCT00490620
Title: Randomized Controlled Pilot Study of Combivir for Patients With Primary Biliary Cirrhosis
Brief Title: Study of Combivir for Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: GlaxoSmithKline (Industry); Axcan Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Col40296
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Primary Biliary Cirrhosis
Keywords: primary biliary cirrhosis C06.552.630.400; retroviral infection C02.782.815
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — lamivudine, zidovudine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): blinded placebo control
  Interventions: Drug: Placebo
- 2 (Active Comparator): Antiretroviral therapy
  Interventions: Drug: Combination antiviral therapy

INTERVENTIONS:
Drug: Combination antiviral therapy — Zidovudine 300mg and lamivudine 150mg BID for 6 months
  Other Names: Combivir
  Arms: 2
Drug: Placebo — placebo BID for 6 months
  Arms: 1

SUMMARY:
This is a proof of principal study to determine whether combination anti-viral therapy with Combivir impacts on hepatic biochemistry in patients with primary biliary cirrhosis

DETAILED DESCRIPTION:
A novel human retrovirus has been cloned from a cDNA library derived from biliary epithelia cells extracted from patients with Primary Biliary Cirrhosis. Although there is no formal proof that this virus is etiologically related to the disease, we have found evidence for viral infection in the majority of patients with PBC using standard serologic and hybridization assays. In order to address the hypotheses that PBC is etiologically related to a retrovirus infection and that anti-retroviral therapy may be beneficial for patients with PBC, we have conducted 2 pilot studies using lamivudine and Combivir (lamivudine 150mg and Zidovudine 300mg). On the whole, little clinical improvement was observed in patients on lamivudine therapy alone, whereas those on Combivir had significant reductions of hepatic biochemistry studies and histologic improvement. Moreover, 4 of 10 Combivir patients completely normalized their liver function tests and the anti-viral therapy was well tolerated. We now propose a larger randomized trial to assess the short term (6 months) safety and efficacy of Combivir for patients with PBC. Efficacy in this study will be defined using both liver biochemistries and virologic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old of either sex will be recruited for this study.
* Persistently elevated alkaline phosphatase or serum aminotransferases of at least 1.5 times normal after a minimum of 6 months UDCA therapy.
* Positive serum AMA (titer > 1:20).
* Liver biopsy histology compatible with PBC obtained at any time prior to study.
* Maintained on UDCA at a dose of 13-15 mg/kg for 6 or more months.
* Patients must read and sign informed consent form.

Exclusion Criteria:

* Patients treated with immunosuppressive or anti-inflammatory agents such as colchicine, methotrexate, D-penicillamine, cyclosporine, tacrolimus, mycophenolate mofetil, corticosteroid therapy will be excluded but may enter the study after a 3 month period off immunosuppressive and anti-inflammatory therapy.
* Advanced liver disease: Childs Pugh class B or C cirrhosis, recurrent variceal hemorrhage, spontaneous encephalopathy, diuretic resistant ascites, need for liver transplantation within the year.
* Patients with a secondary hepatic diagnosis such as viral hepatitis, drug induced liver injury, extrahepatic biliary obstruction, primary sclerosing cholangitis, metabolic liver diseases or alcoholic liver disease.
* Regular use of more than 30 g of alcohol per day in the last year.
* Patients with a predicted survival of less than 3 years from malignant or other potentially life threatening disease.
* Creatinine clearance less than < 70 mL/min using the Cockcroft Gault equation:
* Clinically apparent pancreatitis.
* Serum amylase > 3 x upper limit of normal (patients with sicca syndrome and salivary gland disease may have elevated amylase levels)
* Pregnancy or breast-feeding a child.
* Sexually active patients of child bearing age and not using effective contraception.
* Allergic reaction to Combivir like drugs
* Clinical evidence of myositis
* Weight of < 50 Kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with either (i) normalized alkaline phosphatase, (ii) normalized AST and ALT or (iii) normal alkaline phosphatase, AST and ALT will be recorded. | During the 6 months of therapy

SECONDARY OUTCOMES:
50% improvement towards baseline for alkaline phosphatase, AST and ALT, changes in symptoms using an objective graded clinical parameter scale, serum AMA titers, quantitative immunoglobulins and virologic parameters. | During the 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Mason, MBBS MRCPI, Principal Investigator — University of Alberta; Bruce Bacon, MD, Principal Investigator — St. Louis University; Keith Lindor, MD, Principal Investigator — Mayo Clinic Foundation; James Neuberger, MD FRCP, Principal Investigator — University of Birmingham; Catherine Vincent, MD FRCPC, Principal Investigator — Université de Montréal
Locations (5):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - St Louis University, St Louis, Missouri
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Montreal, Montreal, Quebec
- University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Background] Mason AL, Farr GH, Xu L, Hubscher SG, Neuberger JM. Pilot studies of single and combination antiretroviral therapy in patients with primary biliary cirrhosis. Am J Gastroenterol. 2004 Dec;99(12):2348-55. doi: 10.1111/j.1572-0241.2004.40741.x. PMID 15571581
- [Background] Mason A, Nair S. Primary biliary cirrhosis: new thoughts on pathophysiology and treatment. Curr Gastroenterol Rep. 2002 Feb;4(1):45-51. doi: 10.1007/s11894-002-0037-8. PMID 11825541
- [Background] Xu L, Shen Z, Guo L, Fodera B, Keogh A, Joplin R, O'Donnell B, Aitken J, Carman W, Neuberger J, Mason A. Does a betaretrovirus infection trigger primary biliary cirrhosis? Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8454-9. doi: 10.1073/pnas.1433063100. Epub 2003 Jun 27. PMID 12832623